CLINICAL TRIAL: NCT05902663
Title: Non-interventional Study of Patients With Netherton Syndrome to Characterise the Natural History of Disease
Brief Title: Natural History of Netherton Syndrome
Status: Terminated | Type: Observational
Why Stopped: sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1368-0121; EUPAS103733 (Registry Identifier: EMA RWE catalogues)
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with Netherton Syndrome

SUMMARY:
The goal of this non-interventional study (NIS) is to collect real-world data to describe the natural history of Netherton Syndrome (NS).

ELIGIBILITY:
Inclusion criteria [for Part 1 and Part 2]

1. Confirmed diagnosis of NS by at least one of the following:

   * Genetic testing of mutations in Serine Protease Inhibitor of Kazal Type 5 (SPINK5);
   * Absence or major deficiency of the protein Lympho-Epithelial Kazal-Type-Related Inhibitor (LEKTI) in skin biopsy;
   * Clinical assessment (signs and symptoms).
2. Provision of consent or assent (i.e., by parent or legal guardian) as required by local regulations:

   * [Part 1] to authorise access to existing medical records for study data collection;
   * [Part 2] to participate in the longitudinal 52-week evaluation of disease severity and clinical outcome assessments.

   [for Part 2 only]
3. Not participating in a clinical trial at the time of study enrolment for Part 2.

Exclusion criteria [for Part 1 and Part 2]

1. Patient who has died prior to 2002.
2. Patient whose last known survival status is dated prior to 2002 (i.e., patient has been lost to clinical follow-up since 2002).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sites will identify all patients diagnosed and treated for NS in routine clinical practice to form the base cohort for study eligibility assessment. Patients in the base cohort will be further reviewed for study eligibility based on the criteria below.
  Part 1 - retrospective data collection:
  In Part 1 of the study clinical data will be abstracted from patients' existing medical records from the date of study enrolment back to the date of initial diagnosis of NS.
  Part 2 - prospective data collection:
  In Part 2, patients who are not enrolled in a clinical trial at the time of study inclusion will be asked to provide additional consent/assent to participate in a 52-week follow-up for continuous clinical data collection from medical records and completion of Clinician-Reported Outcomes (ClinRO) and Patient-Reported Outcomes (PRO) assessments.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Severity of Netherton Syndrome (NS) assessed by the Ichthyosis Area Severity Index (IASI) | up to 1 year
  For patients participating in Part 2.
  IASI is a composite score that evaluates severity of erythema (subscale IASI-E) and scaling (subscale IASI-S) in different body regions as a function of their respective body surface areas. Severity of erythema and scaling is rated on a 5-point Likert scale of 0-4 in each of 4 body regions: head and neck (including scalp), arms (including palms), legs (including soles) and trunk, prorated based on body surface area in these body regions and the percentage of involvement in each of these body regions. The total IASI score ranges between 0-48 (i.e., sum of a maximum score of 24 for erythema and maximum score of 24 for scaling). Higher score denotes worse clinical severity.

SECONDARY OUTCOMES:
Severity Netherton Syndrome (NS) assessed by the Investigator Global Assessment (IGA) | up to 1 year
  For patients participating in Part 2.
  IGA for NS will assess the global severity of erythema and scaling in NS using 5-point Likert scale ranging from 0=clear, to 4=severe.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - Northwestern University, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Istituto Dermopatico Dell'Immacolata - IDI - IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com